CLINICAL TRIAL: NCT02255396
Title: Are Estradiol and Testosterone Levels in Seminal Plasma Predictive for Efficient Spermatogenesis in Men With Non- Obstructive Azoospermia
Brief Title: Estradiol and Testosterone Levels in Seminal Plasma of Men With Non-obstructive Azoospermia
Status: Completed | Type: Observational
Sponsor: University Hospital, Clermont-Ferrand (Other)
Responsible Party: Sponsor
Other Study IDs: CHU-209
Record Dates: First submitted 2014-09-26; First posted 2014-10-02 (Estimated); Last update posted 2014-10-02 (Estimated); Status verified 2014-09

CONDITIONS: Non-obstructive Azoospermia With Testicular Biopsy for Spermatozoa Extraction
MeSH Terms: interventions — Estradiol

STUDY DESIGN:
Time Perspective: Cross-Sectional

INTERVENTIONS:
Other: ESTRADIOL

SUMMARY:
Estradiol and Testosterone are two important hormones for the regulation of an effective spermatogenesis in human testis. The evaluation of levels of estradiol and testosterone in seminal plasma of men with non-obstructive azoospermia may be a predictive test before surgical testicular biopsy to determine the chance of a positive sperm extraction to use for ICSI.

DETAILED DESCRIPTION:
The aim of this study is to compare the levels of esttradiol and testosterone in seminal plasma of men with non-obstructive azoospermia. Indeed, for these patients, none biological test allows to predict a positive sperm extraction before the surgical testis biopsy is performed. Since the involvement of estradiol and testosterone in the regulation of spermatogenesis, the measurement of these hormones in seminal plasma may be a predictive tool for these men before testis biopsy.

ELIGIBILITY:
Inclusion Criteria:

* Azoospermia confirmed by two semen analysis (at minimum 74 days between the both analysis)
* Volume of seminal plasma >0.6ml
* Testicular biopsy one month after the last semen analysis
* Informed consent signed by the patient

Exclusion Criteria:

* obstructive azoospermia
* cryptozoospermia

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Study Population: azoospermia
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2009-01; Primary Completion 2013-12 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Levels of estradiol and testosterone in seminal plasma of men with non-obstuctive azoospermia | at 1 month
Issue of testicular biopsy (sperm extraction positive or negative) | at day 1

SECONDARY OUTCOMES:
Degrees of alteration of testis histology | at day 1
Serum levels of estradiol and testosterone | at day 1

CONTACTS AND LOCATIONS:
Locations (1):
- CHU de Clermont-Ferrand, Clermont-Ferrand, France